CLINICAL TRIAL: NCT01668797
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy, Safety, and Tolerability of Brexpiprazole (OPC-34712) as Maintenance Treatment in Adults With Schizophrenia
Brief Title: Efficacy, Safety, and Tolerability of Brexpiprazole (OPC-34712) as Maintenance Treatment in Adults With Schizophrenia
Acronym: EQUATOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 331-10-232; 2011-005766-38 (EudraCT Number)
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Acute Schizophrenia
MeSH Terms: interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo comparator for 52 weeks
  Interventions: Drug: Placebo
- Brexpiprazole (OPC-34712) (Experimental): Brexpiprazole (OPC-34712) for 52 weeks
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Brexpiprazole tablets 1 to 4 mg /day
  Arms: Brexpiprazole (OPC-34712)
Drug: Placebo — Placebo comparator for 52 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of brexpiprazole compared with placebo as maintenance treatment in adults with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a severely debilitating mental illness that affects approximately 1% of the world population. Hallucinations and delusions are the most striking characteristic positive symptoms of schizophrenia; however, more subtle negative symptoms (eg, social withdrawal and lack of emotion, energy, and motivation) may also be present. The first antipsychotics developed for the treatment of schizophrenia were effective against positive symptoms, but showed little efficacy for negative symptoms and were also associated with a high incidence of side effects. Second generation antipsychotics, represent a significant advancement in the treatment of psychotic disorders because they are effective and at the same time exhibit fewer side effects than first generation antipsychotics. Although generally safer than first generation antipsychotics, the second-generation antipsychotics are not devoid of undesirable side effects such as Hyperprolactinemia and weight gain. In addition, the safety of these drugs vary considerably.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years or older to less than 65 years, inclusive (at time of informed consent)
* Subjects with a current diagnosis of schizophrenia, as defined by DSM-IV-TR criteria and a history of the illness for at least three years prior to screening (as per subject, family, healthcare provider, or by previous medical records).
* Subjects with a stable living environment, as demonstrated by the ability to provide contact information for themselves and/or family/friend(s)/caregiver(s).
* Subjects who showed previous response to antipsychotic treatment in the past year.
* Subjects who are currently treated with oral or depot antipsychotics other than clozapine or who have had a recent lapse in antipsychotic treatment requiring chronic treatment with antipsychotic medication for stabilization.
* Subjects who are experiencing a current acute exacerbation of psychotic symptoms requiring stabilization
* Subjects with a history of relapse and/or exacerbation of symptoms when they are not receiving antipsychotic treatment.

Exclusion Criteria:

* Female patients who are breastfeeding or who have a positive pregnancy test (urine) result prior to receiving investigational medicinal product
* Patients presenting a first episode of schizophrenia based on the clinical judgment of the investigator
* Patients who are diagnosed with a disease other than schizophrenia (schizoaffective disorder, major depressive disorder, bipolar disorder, posttraumatic stress disorder, anxiety disorder, delirium, dementia, amnesia, or other cognitive disorder) based on current DSM-IV-TR Axis Ι criteria, or who are diagnosed with a personality disorder (borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial)
* Subjects experiencing acute depressive symptoms within the past 30 days
* Subjects with schizophrenia who are considered resistant/refractory to antipsychotic treatment by history
* Subjects with a significant risk of violent behavior; who represent a risk of committing suicide
* Subjects with clinically significant tardive dyskinesia
* Subjects currently treated with insulin for diabetes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2012-10; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Skuban, M.D., Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (43):
- United States (13):
  - Anaheim, California
  - Cerritos, California
  - Garden Grove, California
  - San Diego, California
  - Tampa, Florida
  - Hoffman Estates, Illinois
  - Saint Charles, Missouri
  - St Louis, Missouri
  - North Platte, Nebraska
  - Las Vegas, Nevada
  - Memphis, Tennessee
  - Dallas, Texas
  - Richmond, Virginia
- Colombia (4):
  - Barranquilla
  - Bello
  - Bogotá
  - Pereira
- Malaysia (4):
  - Kota Bharu, Kelantan
  - Kuala Lumpur, Kuala Lumpur
  - Kajang, Selangor
  - Sabak Bernam
- San Juan, Puerto Rico
- Romania (8):
  - Arad
  - Brasov
  - Bucharest
  - Craiova
  - Focşani
  - Iași
  - Piteşti
  - Târgovişte
- Serbia (4):
  - Belgrade
  - Kragujevac
  - Novi Kneževac
  - Novi Sad
- Turkey (Türkiye) (3):
  - Denizli
  - Diyarbakır
  - Kocaeli
- Ukraine (6):
  - Kharkiv
  - Kherson,Vil. Stepanivka
  - Kyiv
  - Lviv
  - Odesa
  - Simferopol

REFERENCES:
- [Derived] Correll CU, He Y, Therrien F, MacKenzie E, Meehan SR, Weiss C, Hefting N, Hobart M. Effects of Brexpiprazole on Functioning in Patients With Schizophrenia: Post Hoc Analysis of Short- and Long-Term Studies. J Clin Psychiatry. 2022 Mar 1;83(2):20m13793. doi: 10.4088/JCP.20m13793. PMID 35235720
- [Derived] Marder SR, Meehan SR, Weiss C, Chen D, Hobart M, Hefting N. Effects of Brexpiprazole Across Symptom Domains in Patients With Schizophrenia: Post Hoc Analysis of Short- and Long-Term Studies. Schizophr Bull Open. 2021 May 1;2(1):sgab014. doi: 10.1093/schizbullopen/sgab014. eCollection 2021 Jan. PMID 34901863
- [Derived] Correll CU, Shi L, Weiss C, Hobart M, Eramo A, Duffy RA, Weiller E, Baker RA. Successful switching of patients with acute schizophrenia from another antipsychotic to brexpiprazole: comparison of clinicians' choice of cross-titration schedules in a post hoc analysis of a randomized, double-blind, maintenance treatment study. CNS Spectr. 2019 Oct;24(5):507-517. doi: 10.1017/S1092852918001086. PMID 30306884
- [Derived] Fleischhacker WW, Hobart M, Ouyang J, Forbes A, Pfister S, McQuade RD, Carson WH, Sanchez R, Nyilas M, Weiller E. Efficacy and Safety of Brexpiprazole (OPC-34712) as Maintenance Treatment in Adults with Schizophrenia: a Randomized, Double-Blind, Placebo-Controlled Study. Int J Neuropsychopharmacol. 2017 Jan 1;20(1):11-21. doi: 10.1093/ijnp/pyw076. PMID 27566723

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 753 participants were screened at 49 trial sites in the following 7 countries: United States (US, including Puerto Rico), Malaysia, Colombia, Romania, Ukraine, Serbia, and Turkey.
Pre-assignment Details: Trial had Phase A (Conversion) (N= 406), Phase B (Oral Stabilization) (N= 464; 346 rolled over from Phase A and 118 entered directly into Phase B ) and Phase C (Double-Blind Maintenance) with (N= 202 rolled over from Phase B). Participants were randomized in to Phase C in a 1:1 ratio (brexpiprazole:placebo) to receive treatment for up to 52 weeks.
Groups:
- Phase A (Conversion Phase): The purpose of the open-label conversion phase was 2-fold: 1) to cross-titrate the participants current antipsychotic treatment to brexpiprazole monotherapy over a period of 1 to 4 weeks and 2) to allow washout of prohibited medications in preparation for the stabilization phase.
- Phase B (Stabilization Phase): This single-blind stabilization phase was to titrate participants to a dose of brexpiprazole (1 to 4 mg/day) that would maintain stability of psychotic symptoms over 12 consecutive weeks (within a maximum of 36 weeks), while minimizing tolerability issues.
- Phase C - Brexpiprazole (Double-Blind Maintenance Phase): Participants received maintenance treatment daily with brexpiprazole (at the final dose achieved during the stabilization phase) for up to 52 weeks.
- Phase C - Placebo (Double-Blind Maintenance Phase): Participants received placebo orally once daily for 52 weeks.
Period: Phase A (Conversion Phase)
Arm/Group | Phase A (Conversion Phase) | Phase B (Stabilization Phase) | Phase C - Brexpiprazole (Double-Blind Maintenance Phase) | Phase C - Placebo (Double-Blind Maintenance Phase)
Started | 406 | 0 | 0 | 0
Completed | 346 | 0 | 0 | 0
Not Completed | 60 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0
Not completed — Met Withdrawal Criteria | 3 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 16 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 7 | 0 | 0 | 0
Not completed — Adverse Event Without Impending Relapse | 8 | 0 | 0 | 0
Not completed — Terminated Study on Interim Analysis | 19 | 0 | 0 | 0
Period: Phase B (Stabilization Phase)
Arm/Group | Phase A (Conversion Phase) | Phase B (Stabilization Phase) | Phase C - Brexpiprazole (Double-Blind Maintenance Phase) | Phase C - Placebo (Double-Blind Maintenance Phase)
Started | 0 | 464 (N= 464; 346 rolled over from Phase A and 118 entered directly into Phase B) | 0 | 0
Completed | 0 | 202 | 0 | 0
Not Completed | 0 | 262 | 0 | 0
Not completed — Lost to Follow-up | 0 | 16 | 0 | 0
Not completed — Met Withdrawal Criteria | 0 | 22 | 0 | 0
Not completed — Physician Decision | 0 | 11 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 60 | 0 | 0
Not completed — Protocol Violation | 0 | 3 | 0 | 0
Not completed — Lack of Efficacy | 0 | 21 | 0 | 0
Not completed — Adverse Event Without Impending Relapse | 0 | 43 | 0 | 0
Not completed — Terminated Study on Interim Analysis | 0 | 86 | 0 | 0
Period: Phase C (Double-Blind Maintenance Phase)
Arm/Group | Phase A (Conversion Phase) | Phase B (Stabilization Phase) | Phase C - Brexpiprazole (Double-Blind Maintenance Phase) | Phase C - Placebo (Double-Blind Maintenance Phase)
Started | 0 | 0 | 97 (N= 202 rolled over from Phase B) | 105
Completed | 0 | 0 | 14 | 9
Not Completed | 0 | 0 | 83 | 96
Not completed — Lost to Follow-up | 0 | 0 | 4 | 6
Not completed — Met Withdrawal Criteria | 0 | 0 | 3 | 3
Not completed — Physician Decision | 0 | 0 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 5
Not completed — Protocol Violation | 0 | 0 | 2 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 10
Not completed — Lack of Efficacy without AE | 0 | 0 | 11 | 30
Not completed — Adverse Event Without Impending Relapse | 0 | 0 | 4 | 2
Not completed — Terminated Study on Interim Analysis | 0 | 0 | 49 | 38

BASELINE CHARACTERISTICS:
Population: The enrolled sample was defined as all participants who signed the informed consent for the trial and entered Phase A or Phase B.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase C - Brexpiprazole (Double-Blind Maintenance Phase) | Phase C - Placebo (Double-Blind Maintenance Phase) | Total
Number analyzed (Participants) | 97 | 105 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (10.7) | 41.6 (10.6) | 40.2 (10.7)
Gender [Count of Participants; unit: Participants]
  Female | 39 | 40 | 79
  Male | 58 | 65 | 123

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to Exacerbation of Psychotic Symptoms/Impending Relapse in Phase C.
Description: The primary efficacy variable was time to impending relapse from randomization, as assessed by Clinical Global Impression of Improvement (CGI-I) score ≥5, Positive and Negative Syndrome Scale (PANSS) scores for hostility or uncooperativeness ≥5, or ≥20% increase in PANSS Total Score. Impending relapse was defined as meeting any of the following 5 criteria: 1) CGI-I score of ≥ 5 (minimally worse) and increase in individual PANSS items to a score >4 with an absolute increase of ≥ 2 on that specific item or absolute increase of ≥ 4 on the combined 4 PANSS items (conceptual disorganization, hallucinatory behavior, suspiciousness, unusual thought content).OR 2) CGI-I score of 6 or 7 (much or very much worse) OR 3) Hospitalization due to worsening of illness OR 4) Any suicidal behavior or answers of "yes" to Questions 4 or 5 on the suicidal ideation section of the C-SSRS OR 5) Violent or aggressive behavior resulting in clinically significant injury.The measure type, number is Hazard Ratio.
Time Frame: From randomization to time of exacerbation of psychotic symptoms/impending relapse - up to 52 weeks
Population: Based on the Intent-to-Treat (ITT) principle, the full analysis set of this trial was composed of all participants randomized to the double-blind treatment who took at least one dose of study medication in Phase C and who had at least one post-randomization efficacy evaluation in Phase C.
Measure: Number (95% Confidence Interval); unit: Days
Groups:
- Brexpiprazole: Participants received maintenance treatment daily with brexpiprazole (at the final dose achieved during the stabilization phase) for up to 52 weeks.
- Placebo: Participants received placebo orally once daily for 52 weeks.
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Days | 0.292 [0.156 to 0.548] | 3.420 [1.825 to 6.411]
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; The total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 1:1 (brexpiprazole:placebo) randomization ratio; Test type: Superiority or Other; p < 0.0001, Log Rank; The log-rank test was based on time to exacerbation of psychotic symptoms/impending relapse

2. Secondary Outcome: Percentage of Participants Meeting Exacerbation of Psychotic Symptoms/Impending Relapse Criteria in the Double-blind Maintenance Phase
Description: Impending relapse was defined as meeting any of the following 5 criteria: 1) CGI-I score of ≥ 5 (minimally worse) and increase in individual PANSS items to a score > 4 with an absolute increase of ≥ 2 on that specific item or an increase on any of the following individual PANSS items (conceptual disorganization, hallucinatory behavior, suspiciousness, unusual though content) to a score of >4 and an absolute increase of ≥ 4 on the combined 4 PANSS items. OR 2) CGI-I score of 6 or 7 (much or very much worse) OR 3) Hospitalization due to worsening of illness OR 4) Current suicidal behavior as assessed by the C-SSRS (ie, an answer of "yes" to any of the questions on the suicidal behavior section of the C-SSRS 5) Violent or aggressive behavior resulting in clinically significant self-injury to another person, or property damage.
Time Frame: Baseline and Week 52/Early Termination
Population: Based on ITT principle, the full analysis set of this trial was composed of all participants randomized to the double-blind treatment who took at least one dose of study medication in Phase C and who had at least one post-randomization efficacy evaluation in Phase C.
Measure: Number; unit: percentage of participants
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
percentage of participants | 13.54 | 38.46
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; The percentage of participants with impending relapse in treatment groups (Brexpiprazole and placebo) in final analysis for participants meeting at least one of the criteria; Test type: Superiority or Other; p < 0.0001, Chi-squared

3. Other Pre Specified Outcome: Percentage of Participants Meeting Stability Criteria in Double Blind Maintenance Phase
Description: Participants were assessed for stability using the following criteria:1) Outpatient status AND 2) Positive and Negative Syndrome Scale (PANSS) Total Score ≤ 70 AND 3) A score of ≤ 4 (moderate) on each of the following PANSS items (possible scores of 1 to 7 for each item): conceptual disorganization, suspiciousness hallucinatory behavior, unusual thought content, AND 4) Clinical Global Impression - Severity of Illness scale(CGI-S) score ≤ 4 (moderately ill) AND 5) No current suicidal behavior as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS), defined as the following: An answer of "no" to each question on the Suicidal Behavior section of the C-SSRS AND an answer of "no" to Questions 4 and 5 on the Suicidal Ideation section of the C-SSRS, if completed, AND 6) No evidence of aggressive or violent behavior resulting in clinically significant self-injury, injury to another person, property damage.
Time Frame: Weeks 6, 12, 24, 36 and 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
percentage of participants
  Week 6 (N= 81, 84) | 92.59 | 86.90
  Week 12 (N= 73, 68) | 93.15 | 86.76
  Week 24 (N= 50, 36) | 96.00 | 94.44
  Week 36 (N= 33, 24) | 93.94 | 83.33
  Week 52 (N= 15, 9) | 86.67 | 88.89
  Last Visit (N= 96, 104) | 79.17 | 56.73
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.2296, Chi-squared
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.2051, Chi-squared
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.7354, Chi-squared
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.1977, Chi-squared
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.8734, Chi-squared
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Last Visit; Test type: Superiority or Other; p = 0.0007, Chi-squared

4. Other Pre Specified Outcome: Mean Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score - MMRM Analysis
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS total score was the sum of the rating scores for 7 positive scale items, 7 negative scale items, and 16 general psychopathology scale items from the PANSS panel. The PANSS total score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: Based on ITT principle, the full analysis set was composed of all participants randomized to the double-blind treatment who took at least one dose of study medication in Phase C and who had at least one post-randomization efficacy evaluation in Phase C.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 (N= 81, 84) | 0.79 (1.31) | 4.09 (1.27)
  Week 12 (N= 73, 68) | 0.84 (1.73) | 6.15 (1.74)
  Week 24 (N= 50, 36) | -1.88 (1.39) | 2.89 (1.55)
  Week 36 (N= 33, 24) | -2.71 (1.48) | 3.33 (1.70)
  Week 52 (N= 15, 9) | 0.61 (3.34) | 6.92 (4.53)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis of treatment comparisons at Week 6; Test type: Superiority or Other; p = 0.0664, Mixed Models Analysis; Mean Difference (Final Values) = -3.30, 95% CI 2-sided [-6.82 to 0.23]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis of treatment comparisons at Week 12; Test type: Superiority or Other; p = 0.0301, Mixed Models Analysis; Mean Difference (Final Values) = -5.31, 95% CI 2-sided [-10.1 to -0.52]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis of treatment comparisons at Week 24; Test type: Superiority or Other; p = 0.0226, Mixed Models Analysis; Mean Difference (Final Values) = -4.77, 95% CI 2-sided [-8.86 to -0.68]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis of treatment comparisons at Week 36; Test type: Superiority or Other; p = 0.0086, Mixed Models Analysis; Mean Difference (Final Values) = -6.03, 95% CI 2-sided [-10.5 to -1.59]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis of treatment comparisons at Week 52; Test type: Superiority or Other; p = 0.2800, Mixed Models Analysis; Mean Difference (Final Values) = -6.31, 95% CI 2-sided [-18.1 to 5.46]
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Statistical analysis at across visits; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; Mean Difference (Final Values) = -4.42, 95% CI 2-sided [-7.01 to -1.82]

5. Other Pre Specified Outcome: Mean Change From Baseline in PANSS Total Score - Last-observation-carried-forward (LOCF) Analysis
Description: as for outcome 4
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: The LOCF data set for Phase C included data recorded at a given Phase C visit or, if no observation is recorded at that visit, data carried forward from the previous Phase C visit. Baseline data was not be carried forward to impute missing values for the LOCF data set.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 | 0.51 (1.40) | 3.56 (1.28)
  Week 12 | 1.55 (1.77) | 6.60 (1.62)
  Week 24 | 1.58 (1.88) | 9.17 (1.72)
  Week 36 | 2.49 (1.89) | 10.51 (1.73)
  Week 52 | 3.25 (1.94) | 11.20 (1.77)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.0683, ANCOVA; Mean Difference (Final Values) = -3.04, 95% CI 2-sided [-6.31 to 0.23]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.0174, ANCOVA; Mean Difference (Final Values) = -5.05, 95% CI 2-sided [-9.20 to -0.90]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0008, ANCOVA; Mean Difference (Final Values) = -7.59, 95% CI 2-sided [-12.0 to -3.18]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0005, ANCOVA; Mean Difference (Final Values) = -8.02, 95% CI 2-sided [-12.4 to -3.59]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.0007, ANCOVA; Mean Difference (Final Values) = -7.95, 95% CI 2-sided [-12.5 to -3.41]

6. Other Pre Specified Outcome: Mean Change From Baseline in PANSS Positive Subscale Score - MMRM Analysis
Description: PANSS consisted of three subscales: a total of 30 symptom constructs. For each construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS positive subscale score was the sum of the rating scores for the 7 positive scale items from the PANSS panel. The 7 positive symptom constructs are delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. The PANSS positive subscale score ranged from 7 (best possible outcome) to 49 (worst possible outcome).
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 (N= 81, 84) | 0.17 (0.42) | 1.28 (0.41)
  Week 12 (N= 73, 68) | -0.06 (0.50) | 1.81 (0.51)
  Week 24 (N= 50, 36) | -0.84 (0.46) | 0.72 (0.51)
  Week 36 (N= 33, 24) | -0.97 (0.44) | 0.91 (0.51)
  Week 52 (N= 15, 9) | -1.21 (0.73) | 1.50 (0.99)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.0507, Mixed Models Analysis; Mean Difference (Final Values) = -1.11, 95% CI 2-sided [-2.23 to 0.00]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.0080, Mixed Models Analysis; Mean Difference (Final Values) = -1.87, 95% CI 2-sided [-3.24 to -0.50]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0215, Mixed Models Analysis; Mean Difference (Final Values) = -1.56, 95% CI 2-sided [-2.89 to -0.24]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0053, Mixed Models Analysis; Mean Difference (Final Values) = -1.88, 95% CI 2-sided [-3.19 to -0.58]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.339, Mixed Models Analysis; Mean Difference (Final Values) = -2.71, 95% CI 2-sided [-5.20 to -0.22]
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Statistical analysis at across visits; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-2.32 to -0.88]

7. Other Pre Specified Outcome: Mean Change From Baseline in PANSS Positive Subscale Score - LOCF Analysis
Description: as for outcome 6
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 | 0.30 (0.49) | 1.25 (0.45)
  Week 12 | 0.38 (0.59) | 2.24 (0.54)
  Week 24 | 0.49 (0.64) | 3.23 (0.59)
  Week 36 | 0.97 (0.63) | 3.91 (0.58)
  Week 52 | 0.99 (0.64) | 4.17 (0.59)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.1093, ANCOVA; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-2.10 to 0.21]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.0089, ANOVA; Mean Difference (Final Values) = -1.86, 95% CI 2-sided [-3.25 to -0.47]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0005, ANCOVA; Mean Difference (Final Values) = -2.74, 95% CI 2-sided [-4.26 to -1.22]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -2.94, 95% CI 2-sided [-4.43 to -1.44]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -3.18, 95% CI 2-sided [-4.70 to -1.66]

8. Other Pre Specified Outcome: Mean Change From Baseline in PANSS Negative Subscale Score - MMRM Analysis
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS negative subscale score was the sum of the rating scores for the 7 negative scale items from the PANSS panel. The 7 negative symptom constructs: blunted affect, emotional withdrawal, poor rapport, passive apathetic withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. The PANSS negative subscale score ranged from 7 (best possible outcome) to 49 (worst possible outcome).
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 (N= 81, 84) | -0.04 (0.37) | 0.65 (0.35)
  Week 12 (N= 73, 68) | -0.22 (0.43) | 0.55 (0.44)
  Week 24 (N= 50, 36) | -0.78 (0.39) | 0.18 (0.42)
  Week 36 (N= 33, 24) | -1.03 (0.47) | 0.02 (0.53)
  Week 52 (N= 15, 9) | 1.30 (1.37) | 0.87 (1.71)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.1650, Mixed Models Analysis; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-1.66 to 0.29]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.2001, Mixed Models Analysis; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.97 to 0.42]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0939, Mixed Models Analysis; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-2.07 to 0.16]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.1396, Mixed Models Analysis; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-2.44 to 0.35]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.8470, Mixed Models Analysis; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-4.14 to 5.00]
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Statistical analysis at across visits; Test type: Superiority or Other; p = 0.2258, Mixed Models Analysis; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-1.24 to 0.3]

9. Other Pre Specified Outcome: Mean Change From Baseline in PANSS Negative Subscale Score - LOCF Analysis
Description: as for outcome 8
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 | -0.12 (0.39) | 0.63 (0.35)
  Week 12 | -0.17 (0.46) | 1.06 (0.42)
  Week 24 | -0.08 (0.49) | 1.47 (0.44)
  Week 36 | -0.14 (0.51) | 1.44 (0.46)
  Week 52 | 0.39 (0.54) | 1.63 (0.49)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.0981, ANCOVA; Mean Difference (Final Values) = -0.76, 95% CI 2-sided [-1.65 to 0.14]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.0264, ANCOVA; Mean Difference (Final Values) = -1.22, 95% CI 2-sided [-2.30 to -0.15]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0078, ANCOVA; Mean Difference (Final Values) = -1.55, 95% CI 2-sided [-2.69 to -0.42]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0101, ANCOVA; Mean Difference (Final Values) = -1.57, 95% CI 2-sided [-2.77 to -0.38]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.0516, ANCOVA; Mean Difference (Final Values) = -1.24, 95% CI 2-sided [-2.50 to 0.01]

10. Other Pre Specified Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score at Endpoint - MMRM Analysis
Description: The severity of illness for each participant was rated using the CGI-S scale. To assess CGI-S, the study physician answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0 = not assessed; 1 = normal, not ill at all; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Baseline, Weeks 6, 12, 24, 36 and 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 (N= 81, 84) | -0.01 (0.09) | 0.26 (0.09)
  Week 12 (N= 73, 68) | -0.01 (0.11) | 0.37 (0.11)
  Week 24 (N= 50, 36) | -0.16 (0.10) | 0.21 (0.10)
  Week 36 (N= 33, 24) | -0.31 (0.11) | 0.25 (0.12)
  Week 52 (N= 15, 9) | -0.23 (0.17) | 0.28 (0.22)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.0279, Mixed Models Analysis; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.53 to -0.03]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.0117, Mixed Models Analysis; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.68 to -0.09]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0105, Mixed Models Analysis; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.64 to -0.09]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-0.87 to -0.25]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.0780, Mixed Models Analysis; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-1.09 to 0.06]
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Statistical analysis at across visits; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.54 to -0.15]

11. Other Pre Specified Outcome: Change From Baseline in CGI-S Score at Endpoint - LOCF Analysis
Description: as for outcome 10
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 | -0.08 (0.09) | 0.17 (0.09)
  Week 12 | -0.04 (0.11) | 0.32 (0.10)
  Week 24 | -0.03 (0.11) | 0.47 (0.10)
  Week 36 | -0.00 (0.11) | 0.56 (0.10)
  Week 52 | 0.02 (0.11) | 0.55 (0.11)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.0284, ANCOVA; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.47 to -0.03]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.0056, ANCOVA; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.62 to -0.11]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.76 to -0.24]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-0.82 to -0.30]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-0.79 to -0.26]

12. Other Pre Specified Outcome: Clinical Global Impression - Improvement Score (CGI-I) at Endpoint - LOCF Analysis
Description: The rater or investigator would rate the participant's total improvement whether or not it is due entirely to study treatment. During Phase B, responses were compared to the participant's condition at Baseline of Phase B (for participants who entered Phase B directly after screening) or to the End of Phase A visit (for participants who participated in Phase A). During Phase C, responses were compared to the participant's condition at the End of Phase B visit. Response choices include: 0 = Not assessed, 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, and 7 = Very much worse.
Time Frame: Weeks 6, 12, 24, 36 and 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 | 3.68 (0.98) | 4.00 (1.14)
  Week 12 | 3.66 (1.19) | 4.10 (1.30)
  Week 24 | 3.67 (1.27) | 4.30 (1.32)
  Week 36 | 3.71 (1.27) | 4.39 (1.30)
  Week 52 | 3.77 (1.26) | 4.40 (1.32)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.0387, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.60 to -0.20]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.0185, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.75 to -0.07]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0010, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.97 to -0.24]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0004, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-1.02 to -0.30]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel; Treatment difference = -0.61, 95% CI 2-sided [-0.96 to -0.25]

13. Other Pre Specified Outcome: Mean Change From Baseline in Personal and Social Performance (PSP) Scale Score - MMRM Analysis
Description: The PSP is a validated clinician-rated scale that measures personal and social functioning in four domains: socially useful activities (e.g., work and study), personal and social relationships, self-care, and disturbing and aggressive behaviors. Impairment in each of these domains is rated as absent, mild, manifest, marked, severe, or very severe. These ratings are then converted to a total score based on a 100-point scale using algorithms to identify the appropriate 10-point interval, and the rater's judgment to determine the total score within the 10-point interval. Participants with a PSP total score of 71 to 100 are considered to have mild functional difficulty. Scores of 31 to 70 represent manifest disabilities of various degrees and ratings of 1 to 30 indicate minimal functioning that requires intense support and/or supervision.The PSP score ranges from 0 to 100, with higher scores indicating higher levels of social functioning.
Time Frame: Baseline and Weeks 24 and 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 24 (N= 50, 36) | 18.85 (1.51) | 17.84 (1.82)
  Week 52 (N= 15, 9) | 18.63 (2.76) | 12.55 (3.48)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.6525, Mixed Models Analysis; Mean Difference (Final Values) = 1.01, 95% CI 2-sided [-3.47 to 5.49]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.1677, Mixed Models Analysis; Mean Difference (Final Values) = 6.08, 95% CI 2-sided [-2.71 to 14.87]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at across visits; Test type: Superiority or Other; p = 0.2347, Mixed Models Analysis; Mean Difference (Final Values) = 3.55, 95% CI 2-sided [-2.41 to 9.5]

14. Other Pre Specified Outcome: Mean Change From Baseline in PSP Scale Score - LOCF Analysis
Description: as for outcome 13
Time Frame: Baseline and Weeks 24 and 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 94 | 100
Units on a scale
  Week 24 | 15.20 (1.41) | 11.41 (1.32)
  Week 52 | 15.06 (1.43) | 10.31 (1.34)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0285, ANCOVA; Mean Difference (Final Values) = 3.79, 95% CI 2-sided [0.40 to 7.17]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.0071, ANCOVA; Mean Difference (Final Values) = 4.75, 95% CI 2-sided [1.31 to 8.18]

15. Other Pre Specified Outcome: Mean Change From Baseline in Global Assessment of Functioning (GAF) Scale Score - MMRM Analysis
Description: The GAF is a clinician-rated scale that assesses the participant's psychological, social, and occupational functioning on a hypothetical continuum of mental health-illness using a scale that ranges from 1 to 100 score, where lower values indicate worst outcome. From among 10 descriptive anchors, investigators will choose the anchor which is the most representative of the participant's level of functioning at the time of the assessment and will assign a single score within the point range given for the selected anchor.
Time Frame: Baseline and Weeks 12, 24, 36 and 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 12 (N= 73, 68) | 1.59 (1.27) | -0.03 (1.29)
  Week 24 (N= 50, 36) | 3.74 (1.42) | 1.09 (1.57)
  Week 36 (N= 33, 24) | 4.71 (1.50) | 0.21 (1.67)
  Week 52 (N= 15, 9) | 5.72 (1.87) | -0.16 (2.37)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.3290, Mixed Models Analysis; Mean Difference (Final Values) = 1.61, 95% CI 2-sided [-1.65 to 4.88]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.1765, Mixed Models Analysis; Mean Difference (Final Values) = 2.66, 95% CI 2-sided [-1.22 to 6.54]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0331, Mixed Models Analysis; Mean Difference (Final Values) = 4.50, 95% CI 2-sided [0.38 to 8.63]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.0522, Mixed Models Analysis; Mean Difference (Final Values) = 5.88, 95% CI 2-sided [-0.06 to 11.82]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at across visits; Test type: Superiority or Other; p = 0.0281, Mixed Models Analysis; Mean Difference (Final Values) = 3.66, 95% CI 2-sided [0.41 to 6.92]

16. Other Pre Specified Outcome: Mean Change From Baseline in GAF Scale Score - LOCF Analysis
Description: as for outcome 15
Time Frame: Baseline and Weeks 12, 24, 36 and 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 95 | 102
Units on a scale
  Week 12 | 0.44 (1.26) | -3.44 (1.17)
  Week 24 | 0.85 (1.37) | -4.51 (1.27)
  Week 36 | 0.97 (1.35) | -5.84 (1.25)
  Week 52 | 0.55 (1.38) | -6.01 (1.28)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.0111, ANCOVA; Mean Difference (Final Values) = 3.88, 95% CI 2-sided [0.90 to 6.86]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0014, ANCOVA; Mean Difference (Final Values) = 5.36, 95% CI 2-sided [2.10 to 8.62]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Final Values) = 6.81, 95% CI 2-sided [3.61 to 10.00]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = 6.55, 95% CI 2-sided [3.28 to 9.83]

17. Other Pre Specified Outcome: Percentage of Participants Who Discontinued Due to All Causes
Description: Analysis of the percentage of participants who discontinued due to all causes was based on all participants who have been randomized and taken one dose of IMP in the Double-blind Maintenance phase. The trial was completed by sponsor when efficacy was demonstrated at the first pre-specified interim analysis (45 impending relapse events) performed by an independent (unblinded) statistician.
Time Frame: Baseline to Week 52
Population: as for outcome 4
Measure: Number; unit: Percentage of particpants
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Percentage of particpants | 34.38 | 54.81
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Test type: Superiority or Other; p = 0.0014, Log Rank

18. Other Pre Specified Outcome: Mean Change From Baseline in PANSS Excited Component (PEC) Score - MMRM Analysis
Description: The PEC score consisted of five PANSS items: excitement (P4), hostility (P7), tension (G4), uncooperativeness (G8), and poor impulse control (G14). Each of the items were rated on a scale of 1 (absent) to 7 (extreme). The PEC scores ranged from 5 (not present) to 35 (extremely severe).
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: The last-observation-carried-forward (LOCF) data set included data recorded at a given Phase C visit or, if no observation is recorded at that visit, data carried forward from the previous Phase C visit. Baseline data (eg.the last visit prior to the first dosing of Phase C) were not be carried forward to impute missing values for the LOCF data set.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 (N= 81, 84) | 0.32 (0.23) | 0.74 (0.22)
  Week 12 (N= 73, 68) | 0.50 (0.34) | 1.16 (0.35)
  Week 24 (N= 50, 36) | -0.06 (0.31) | 0.45 (0.36)
  Week 36 (N= 33, 24) | 0.10 (0.33) | 1.25 (0.40)
  Week 52 (N= 15, 9) | -0.04 (0.46) | 1.00 (0.59)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.1577, Mixed Models Analysis; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-1.02 to 0.17]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.1685, Mixed Models Analysis; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-1.61 to 0.28]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.2815, Mixed Models Analysis; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.43 to 0.42]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0286, Mixed Models Analysis; Mean Difference (Final Values) = -1.14, 95% CI 2-sided [-2.16 to -0.12]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.1803, Mixed Models Analysis; Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-2.58 to 0.51]
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Statistical analysis at across visits; Test type: Superiority or Other; p = 0.0077, Mixed Models Analysis; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-1.12 to -0.17]

19. Other Pre Specified Outcome: Mean Change From Baseline in PEC Score - LOCF Analysis
Description: as for outcome 18
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 | 0.38 (0.27) | 0.81 (0.25)
  Week 12 | 0.73 (0.36) | 1.36 (0.33)
  Week 24 | 0.78 (0.42) | 1.86 (0.38)
  Week 36 | 0.89 (0.41) | 2.23 (0.38)
  Week 52 | 0.82 (0.41) | 2.35 (0.38)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.1852, ANCOVA; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.06 to 0.21]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.1430, ANCOVA; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-1.47 to 0.21]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0323, ANCOVA; Mean Difference (Final Values) = -1.08, 95% CI 2-sided [-2.06 to -0.09]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0071, ANCOVA; Mean Difference (Final Values) = -1.34, 95% CI 2-sided [-2.31 to -0.37]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.0023, ANCOVA; Mean Difference (Final Values) = -1.54, 95% CI 2-sided [-2.52 to -0.56]

20. Other Pre Specified Outcome: Mean Change From Baseline in PANSS Marder Factor Scores: Positive Symptoms Score - MMRM Analysis
Description: Retrospective factor analyses have been performed in recent decades using scores for the 30 individual PANSS items to categorize symptoms into 5 dimensions. Collectively, these dimensions are referred to as the PANSS Marder Factor scores and include positive symptoms score, negative symptoms score, thought score, uncontrolled hostility/excitement, anxiety depression score. The positive factor score is the sum of the 8 components of the positive symptoms scale (range: 8 - best possible outcome to 56 - worst possible outcome).
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 (N= 81, 84) | -0.10 (0.45) | 1.24 (0.44)
  Week 12 (N= 73, 68) | -0.18 (0.58) | 1.83 (0.58)
  Week 24 (N= 50, 36) | -0.82 (0.54) | 0.77 (0.60)
  Week 36 (N= 33, 24) | -1.35 (0.57) | 0.93 (0.63)
  Week 52 (N= 15, 9) | -1.62 (0.83) | 1.78 (1.05)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.0288, Mixed Models Analysis; Mean Difference (Final Values) = -1.34, 95% CI 2-sided [-2.54 to -0.14]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.0128, Mixed Models Analysis; Mean Difference (Final Values) = -2.02, 95% CI 2-sided [-3.60 to -0.44]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0462, Mixed Models Analysis; Mean Difference (Final Values) = -1.59, 95% CI 2-sided [-3.15 to 0.03]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0074, Mixed Models Analysis; Mean Difference (Final Values) = -2.29, 95% CI 2-sided [-3.94 to -0.64]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.0136, Mixed Models Analysis; Mean Difference (Final Values) = -3.40, 95% CI 2-sided [-6.05 to -0.75]
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Statistical analysis at across visits; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.91, 95% CI 2-sided [-2.84 to -0.97]

21. Other Pre Specified Outcome: Mean Change From Baseline in PANSS Marder Factor Scores: Positive Symptoms Score - LOCF Analysis
Description: as for outcome 20
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 | 0.05 (0.50) | 1.13 (0.46)
  Week 12 | 0.10 (0.61) | 2.03 (0.56)
  Week 24 | 0.25 (0.66) | 3.08 (0.61)
  Week 36 | 0.60 (0.66) | 3.69 (0.60)
  Week 52 | 0.58 (0.66) | 4.02 (0.60)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.0695, ANCOVA; Mean Difference (Final Values) = -1.08, 95% CI 2-sided [-2.26 to 0.09]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.0089, ANCOVA; Mean Difference (Final Values) = -1.93, 95% CI 2-sided [-3.38 to -0.49]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0004, ANCOVA; Mean Difference (Final Values) = -2.83, 95% CI 2-sided [-4.39 to -1.27]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -3.09, 95% CI 2-sided [-4.63 to -1.54]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -3.44, 95% CI 2-sided [-4.99 to -1.89]

22. Other Pre Specified Outcome: Mean Change From Baseline in PANSS Marder Factor Scores: Negative Symptoms Score - MMRM Analysis
Description: Retrospective factor analyses have been performed in recent decades using scores for the 30 individual PANSS items to categorize symptoms into 5 dimensions. Collectively, these dimensions are referred to as the PANSS Marder Factor scores and include positive symptoms score, negative symptoms score, thought score, uncontrolled hostility/excitement, anxiety depression score. The negative factor score is the sum of the 7 items of the negative subscale (range: 8 - best possible outcome to 56 - worst possible outcome).
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 (N= 81, 84) | 0.02 (0.38) | 0.68 (0.36)
  Week 12 (N= 73, 68) | -0.01 (0.45) | 0.80 (0.45)
  Week 24 (N= 50, 36) | -0.71 (0.40) | 0.46 (0.43)
  Week 36 (N= 33, 24) | -0.80 (0.50) | 0.70 (0.56)
  Week 52 (N= 15, 9) | 1.37 (1.39) | 1.06 (1.77)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.1969, Mixed Models Analysis; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-1.66 to 0.35]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.2007, Mixed Models Analysis; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-2.04 to 0.43]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0436, Mixed Models Analysis; Mean Difference (Final Values) = -1.17, 95% CI 2-sided [-2.30 to -0.03]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0444, Mixed Models Analysis; Mean Difference (Final Values) = -1.51, 95% CI 2-sided [-2.97 to -0.04]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.8927, Mixed Models Analysis; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-4.40 to 5.02]
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Statistical analysis at across visits; Test type: Superiority or Other; p = 0.2154, Mixed Models Analysis; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.34 to 0.31]

23. Other Pre Specified Outcome: Mean Change From Baseline in PANSS Marder Factor Scores: Negative Symptoms Score - LOCF Analysis
Description: as for outcome 22
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 | -0.24 (0.40) | 0.61 (0.36)
  Week 12 | -0.15 (0.48) | 1.09 (0.43)
  Week 24 | -0.09 (0.49) | 1.50 (0.44)
  Week 36 | -0.07 (0.52) | 1.56 (0.47)
  Week 52 | 0.34 (0.56) | 1.57 (0.50)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.0707, ANCOVA; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-1.78 to 0.07]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.0276, ANCOVA; Mean Difference (Final Values) = -1.24, 95% CI 2-sided [-2.35 to -0.14]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0065, ANCOVA; Mean Difference (Final Values) = -1.59, 95% CI 2-sided [-2.72 to -0.45]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0085, ANCOVA; Mean Difference (Final Values) = -1.63, 95% CI 2-sided [-2.84 to -0.42]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.0630, ANCOVA; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-2.52 to 0.07]

24. Other Pre Specified Outcome: Mean Change From Baseline in PANSS Marder Factor Scores: Disorganized Thought Score - MMRM Analysis
Description: Retrospective factor analyses have been performed in recent decades using scores for the 30 individual PANSS items to categorize symptoms into 5 dimensions. Collectively, these dimensions are referred to as the PANSS Marder Factor scores and include positive symptoms score, negative symptoms score, thought score, uncontrolled hostility/excitement, anxiety depression score. The disorganized thoughts factor score is the sum of score from the 7 items on the disorganized thoughts subscale (range: 7 - best possible outcome to 49 - worst possible outcome).
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 (N= 81, 84) | -0.18 (0.31) | 0.32 (0.30)
  Week 12 (N= 73, 68) | -0.44 (0.38) | 0.69 (0.39)
  Week 24 (N= 50, 36) | -1.26 (0.34) | 0.27 (0.38)
  Week 36 (N= 33, 24) | -1.31 (0.44) | 0.17 (0.50)
  Week 52 (N= 15, 9) | -0.37 (0.99) | -0.30 (1.24)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.2251, Mixed Models Analysis; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-1.33 to 0.31]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.0368, Mixed Models Analysis; Mean Difference (Final Values) = -1.13, 95% CI 2-sided [-2.19 to -0.07]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0024, Mixed Models Analysis; Mean Difference (Final Values) = -1.53, 95% CI 2-sided [-2.51 to -0.56]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0293, Mixed Models Analysis; Mean Difference (Final Values) = -1.48, 95% CI 2-sided [-2.80 to -0.15]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.9632, Mixed Models Analysis; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-3.32 to 3.17]
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Statistical analysis at across visits; Test type: Superiority or Other; p = 0.0029, Mixed Models Analysis; Mean Difference (Final Values) = -0.99, 95% CI 2-sided [-1.63 to -0.34]

25. Other Pre Specified Outcome: Mean Change From Baseline in PANSS Marder Factor Scores: Disorganized Thought Score - LOCF Analysis
Description: as for outcome 24
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 | -0.32 (0.34) | 0.33 (0.31)
  Week 12 | -0.19 (0.41) | 1.19 (0.38)
  Week 24 | -0.29 (0.44) | 1.76 (0.41)
  Week 36 | 0.00 (0.45) | 1.95 (0.42)
  Week 52 | 0.29 (0.48) | 1.97 (0.45)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.1062, ANCOVA; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-1.44 to 0.14]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.0051, ANCOVA; Mean Difference (Final Values) = -1.37, 95% CI 2-sided [-2.33 to -0.42]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -2.05, 95% CI 2-sided [-3.08 to -1.01]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0004, ANCOVA; Mean Difference (Final Values) = -1.94, 95% CI 2-sided [-3.00 to -0.89]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.0035, ANCOVA; Mean Difference (Final Values) = -1.69, 95% CI 2-sided [-2.81 to -0.56]

26. Other Pre Specified Outcome: Mean Change From Baseline in PANSS Marder Factor Scores: Uncontrolled Hostility/Excitement Score - MMRM Analysis
Description: Retrospective factor analyses have been performed in recent decades using scores for the 30 individual PANSS items to categorize symptoms into 5 dimensions. Collectively, these dimensions are referred to as the PANSS Marder Factor scores and include positive symptoms score, negative symptoms score, thought score, uncontrolled hostility/excitement, anxiety depression score. The uncontrolled hostility/excitement factor score is the sum of score from the 4 items on the uncontrolled hostility/excitement subscale (range: 4 - best possible outcome to 28 - worst possible outcome).
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 (N= 81, 84) | 0.19 (0.19) | 0.55 (0.18)
  Week 12 (N= 73, 68) | 0.33 (0.28) | 0.82 (0.29)
  Week 24 (N= 50, 36) | -0.26 (0.27) | 0.81 (0.31)
  Week 36 (N= 33, 24) | -0.13 (0.29) | 0.94 (0.34)
  Week 52 (N= 15, 9) | -0.20 (0.40) | 0.94 (0.50)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.1465, Mixed Models Analysis; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.85 to 0.13]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.2154, Mixed Models Analysis; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.27 to 0.29]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.2696, Mixed Models Analysis; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-1.23 to 0.35]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0179, Mixed Models Analysis; Mean Difference (Final Values) = -1.07, 95% CI 2-sided [-1.95 to -0.19]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.0875, Mixed Models Analysis; Mean Difference (Final Values) = -1.14, 95% CI 2-sided [-2.46 to 0.18]
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Statistical analysis at across visits; Test type: Superiority or Other; p = 0.0021, Mixed Models Analysis; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-1.08 to -0.24]

27. Other Pre Specified Outcome: Mean Change From Baseline in PANSS Marder Factor Scores: Uncontrolled Hostility/Excitement Score - LOCF Analysis
Description: as for outcome 26
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 | 0.32 (0.22) | 0.65 (0.21)
  Week 12 | 0.52 (0.30) | 0.94 (0.28)
  Week 24 | 0.50 (0.36) | 1.31 (0.33)
  Week 36 | 0.57 (0.36) | 1.63 (0.33)
  Week 52 | 0.49 (0.37) | 1.75 (0.34)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.2135, ANCOVA; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.86 to 0.19]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.2437, ANCOVA; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.13 to 0.29]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0635, ANCOVA; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.66 to 0.05]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0144, ANCOVA; Mean Difference (Final Values) = -1.07, 95% CI 2-sided [-1.92 to -0.22]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.0046, ANCOVA; Mean Difference (Final Values) = -1.26, 95% CI 2-sided [-2.12 to -0.39]

28. Other Pre Specified Outcome: Mean Change From Baseline in PANSS Marder Factor Scores: Anxiety/Depression Score - MMRM Analysis
Description: Retrospective factor analyses have been performed in recent decades using scores for the 30 individual PANSS items to categorize symptoms into 5 dimensions. Collectively, these dimensions are referred to as the PANSS Marder Factor scores and include positive symptoms score, negative symptoms score, thought score, uncontrolled hostility/excitement, anxiety depression score. The anxiety/depression factor score is the sum of score from the 4 items on the anxiety/depression subscale (range: 4 - best possible outcome to 28 - worst possible outcome).
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 (N= 81, 84) | 0.19 (0.25) | 0.66 (0.24)
  Week 12 (N= 73, 68) | 0.54 (0.29) | 0.78 (0.29)
  Week 24 (N= 50, 36) | 0.61 (0.28) | 0.58 (0.32)
  Week 36 (N= 33, 24) | 0.46 (0.33) | 0.71 (0.39)
  Week 52 (N= 15, 9) | 0.04 (0.43) | 0.28 (0.56)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.1640, Mixed Models Analysis; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-1.14 to 0.19]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.5466, Mixed Models Analysis; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-1.04 to 0.55]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.9417, Mixed Models Analysis; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.81 to 0.87]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.6257, Mixed Models Analysis; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-1.25 to 0.76]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.7437, Mixed Models Analysis; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-1.68 to 1.21]
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Statistical analysis at across visits; Test type: Superiority or Other; p = 0.4506, Mixed Models Analysis; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.62 to 0.28]

29. Other Pre Specified Outcome: Mean Change From Baseline in PANSS Marder Factor Scores: Anxiety/Depression Score - LOCF Analysis
Description: as for outcome 28
Time Frame: Baseline and Weeks 6, 12, 24, 36 and 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 96 | 104
Units on a scale
  Week 6 | 0.19 (0.27) | 0.85 (0.25)
  Week 12 | 0.86 (0.32) | 1.41 (0.30)
  Week 24 | 1.07 (0.32) | 1.64 (0.30)
  Week 36 | 1.09 (0.32) | 1.79 (0.30)
  Week 52 | 1.17 (0.31) | 1.88 (0.29)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.0467, ANCOVA; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-1.32 to -0.06]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.1599, ANCOVA; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-1.33 to 0.22]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.1417, ANCOVA; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-1.35 to 0.19]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0724, ANCOVA; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.47 to 0.06]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Statistical analysis at Week 52; Test type: Superiority or Other; p = 0.0608, ANCOVA; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-1.47 to 0.03]

ADVERSE EVENTS:
Time Frame: Adverse events reported from the signing of the informed consent throughout the stabilization and treatment period followed by a follow-up phone call or clinic visit (study physician's discretion) of 30 (+2) days after last dose of study medication.
Description: AEs were collected for participants who received brexpiprazole in the stabilization phase and for participants were randomized to double-blind treatment (brexpiprazole or placebo) and received at least one dose of double-blind study medication in Double-Blind Maintenance Phase.
Groups:
- Single Blind Stabilization Phase: This single-blind stabilization phase was to titrate participants to a dose of brexpiprazole (1 to 4 mg/day) that would maintain stability of psychotic symptoms over 12 consecutive weeks (within a maximum of 36 weeks), while minimizing tolerability issues.
- Brexpiprazole (Double-blind Maintenance Phase): Participants received maintenance treatment daily with brexpiprazole (at the final dose achieved during the stabilization phase) for up to 52 weeks.
- Placebo (Double-blnd Maintenance Phase): Participants received placebo orally once daily for 52 weeks.
Arm/Group | Single Blind Stabilization Phase | Brexpiprazole (Double-blind Maintenance Phase) | Placebo (Double-blnd Maintenance Phase)
Serious Adverse Events (participants affected / at risk) | 34/464 | 3/97 | 11/104
Other Adverse Events (participants affected / at risk) | 148/464 | 0/97 | 0/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Blind Stabilization Phase (N=464) | Brexpiprazole (Double-blind Maintenance Phase) (N=97) | Placebo (Double-blnd Maintenance Phase) (N=104)
Angina unstable (Cardiac disorders) | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 4
Schizophrenia (Psychiatric disorders) | 22 | 1 | 5
Suicidal ideation (Psychiatric disorders) | 3 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 3 | 0 | 0
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Blind Stabilization Phase (N=464) | Brexpiprazole (Double-blind Maintenance Phase) (N=97) | Placebo (Double-blnd Maintenance Phase) (N=104)
Weight increased (Investigations) | 24 | 0 | 0
Akathisia (Nervous system disorders) | 42 | 0 | 0
Headache (Nervous system disorders) | 23 | 0 | 0
Agitation (Psychiatric disorders) | 30 | 0 | 0
Insomnia (Nervous system disorders) | 56 | 0 | 0
Schizophrenia (Nervous system disorders) | 28 | 0 | 0

LIMITATIONS AND CAVEATS:
As the interim analysis results were positive, the trial was completed as it achieved the primary endpoint of a significant delay in time to impending relapse for participants randomized to brexpiprazole when compared to participants in placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No